CLINICAL TRIAL: NCT00201266
Title: Histoblood Group Antigens, Viruses and Asthma
Brief Title: Histoblood Group Antigens as a Risk Factor of Asthma
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 283; R01HL080414 (NIH)
Record Dates: First submitted 2005-09-16; First posted 2005-09-20 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases | interventions — Mass Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, plasma, saliva, induced sputum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exacerbation resistant asthma: Control group
  Interventions: Procedure: Screening
- Exacerbation prone asthma: Cases
  Interventions: Procedure: Screening

INTERVENTIONS:
Procedure: Screening — Characterization tests including blood group typing, measures of lung function, measures of allergy, and collection of DNA.

SUMMARY:
This study will evaluate the link between blood group antigens and asthma exacerbations.

DETAILED DESCRIPTION:
BACKGROUND:

The purpose of this study is to explore the role of histoblood group antigens in virus-induced asthma exacerbations. These antigens (ABH and Lewis) decorate O- and N-linked glycans on mucin and epithelial glycoproteins, respectively. Glycan synthesis involves glycosyltransferases, including fucosyltransferases (FUT) encoded by FUT genes. Glycan degradation involves glycosidases, including fucosidase. "Secretor status" is defined by FUT2 activity in epithelial cells, which forms the H antigen and allows subsequent synthesis and secretion of A, B, and Lewis B antigens. In preliminary studies it was found that: 1) asthmatic patients with frequent exacerbations are more likely than non-exacerbated patients to be secretors; 2) secretors report more frequently that a cold causes asthma; and 3) sputum in stable asthma has abnormally high fucosidase activity. These findings suggest that airway glycans are subjected to the following two competing homoeostatic influences: 1) the diversity and activity of glycosyltransferases within cells that synthesize glycans; and 2) the diversity and activity of glycosidases that turn over and remodel glycans in the airway lumen. This study will test the hypothesis that secretor positive asthmatic patients are susceptible to virus-induced asthma exacerbation and that abnormal glycosidase activity in secretions modifies the glycan coat and promotes virus-induced exacerbation.

DESIGN NARRATIVE:

Secretor status will be studied in order to determine whether it is a risk factor for asthma exacerbations precipitated by viruses. Preliminary studies suggest that secretor positive asthmatics are prone to asthma exacerbations and that asthmatic patients have abnormal glycosidase activity in their airway secretions. This study will explore these findings further in the following two ways: 1) a case-control study will compare secretor status and frequency of viral airway infection in 50 asthmatic patients hospitalized for management of acute severe asthma to 50 asthmatic subjects in the outpatient setting without a history of severe asthma exacerbation. Sputum samples or tracheal aspirates (from intubated patients) will be collected from all patients. In these samples, DNA will be used as a microarray to detect viruses; and 2) epithelial brushings and bronchial biopsies from a tissue bank will be used to establish the relationship between secretor status (erythrocyte Lea and Leb phenotyping) and airway epithelial cell activity of FUT genes (real time RT-PCR), and expression of Lea, Leb, A, B, and H antigens (immunohistochemistry).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of asthma, as confirmed by methacholine responsiveness less than 8 mg/mL
* History of asthma exacerbation in the 2 years prior to study entry requiring treatment with oral corticosteroids

Exclusion Criteria:

* Cigarette smoking in the 10 years prior to study entry or total pack per year history greater than 10
* History of asthma exacerbations requiring treatment with oral corticosteroids since age 12 (control group)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthmatics of two types: 1. Exacerbation resistant asthma (no requirement for prednisone for asthma since age 12). 2. Exacerbation prone asthma (requirement for prednisone for asthma in the past 2 years).
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2005-07; Primary Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Asthma exacerbations requiring prednisone | Prior 2 years

SECONDARY OUTCOMES:
Lung fuction | Current
  FEV1% predicted

CONTACTS AND LOCATIONS:
Overall Officials: John V. Fahy, Study Chair — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Derived] Innes AL, McGrath KW, Dougherty RH, McCulloch CE, Woodruff PG, Seibold MA, Okamoto KS, Ingmundson KJ, Solon MC, Carrington SD, Fahy JV. The H antigen at epithelial surfaces is associated with susceptibility to asthma exacerbation. Am J Respir Crit Care Med. 2011 Jan 15;183(2):189-94. doi: 10.1164/rccm.201003-0488OC. Epub 2010 Aug 23. PMID 20732988